CLINICAL TRIAL: NCT01291472
Title: Disposition of Intravenous Ketorolac After Cesarean Section
Brief Title: Disposition of Intravenous Ketorolac
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3214; 2011-000367-27 (EudraCT Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-08 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-02

CONDITIONS: Postoperative Pain
Keywords: ketorolac; pain; pregnancy; non-pregnant state
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ketorolac (Other): Ketorolac will be given to all patients as a part of routine medical care
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — After dilution (solution for injection, 10 mg/1ml) in 50-100 ml bag of normal saline drug will be administered by iv bolus, through a peripherally inserted venous catheter, 30 mg, 3 times in one day. The intended duration of administration is 5-10 minutes.
  Other Names: Taradyl

SUMMARY:
The purpose of this study is:

* to document ketorolac disposition (concentration/time profile, protein binding, metabolism) and its covariates following intravenous (iv) administration of ketorolac right after caesarean section and to compare those observations (n=32) with non-pregnant state (n=8) (intra-subject PK comparison)
* to document biochemical tolerance of ketorolac
* to evaluate if optimalisation of ketorolac dose regimen during pregnancy and labor are appropriated and needed
* to quantify the neonatal exposure to ketorolac through excretion in the breast milk

DETAILED DESCRIPTION:
Prospective, single-center, open label study on the pharmacokinetics of intravenous (iv) ketorolac administration in pregnant women right after caesarean section. Patients will be included after signed informed consent. Ketorolac has been selected for this study as it is routinely administered for postoperative pain relief. At this stage, we only have the intention to document ketorolac pharmacokinetics and metabolism based on the dosing regimen as currently used in the clinical setting, and therefore will not interfere with either clinical indications, nor with dosing as prescribed by the attending physician. This drug is routinely administered (30 mg q8h) after caesarean section.

Drug administration and collection of samples will be obtained to the current clinical and nursing standard procedures. After dilution in 50-100 ml bag of normal saline drug will be administered after caesarean section by iv bolus, through a peripherally inserted venous catheter, 30 mg, 3 times in one day. The intended duration of administration is 5-10 minutes.

Blood samples will be collected (in heparinised tubes) according to following schedule: 1, 2, 3, 4, 6 and 8 hours after iv administration, through a second peripherally inserted venous catheter dedicated for blood sampling only. Blood samples will be centrifuged immediately after collection and subsequently stored at -20 °C until analysis. Urine samples will also be collected, before drug administration in the first 8 hours after the first drug administration, through a bladder catheter in patients in whom a bladder catheter is available for clinical indications.

In a subgroup of former patients (n=8), we plan to repeat this procedure 6-12 weeks after delivery (for intra-subject PK comparison). However, only a single iv ketorolac dose will be administered, and sampling will be limited to 6 samples up to 8 h following start of iv administration. A population pharmacokinetics approach will be used, hereby comparing the data on PK already reported in adults and the newly collected data following pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* signed informed written consent
* pregnant women to whom ketorolac is administered by intravenous route for clinical indications
* preferable availability for revision in 6-12 weeks after delivery (around routine post-delivery check-up).

Exclusion Criteria:

* withdrawal of informed written consent
* known NSAID's intolerance

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
ketorolac disposition following intravenous administration right after caesarean section | up to 8 hours after first dose administration
  PK (concentration/time profile, protein binding, metabolism) and its covariates

SECONDARY OUTCOMES:
optimalisation of ketorolac dose regimen during pregnancy and labor | up to 8 hours after first dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Karel Allegaert, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Kulo A, Hendrickx S, de Hoon J, Mulabegovic N, van Calsteren K, Verbesselt R, Allegaert K. The impact of pregnancy on urinary ketorolac metabolites after single intravenous bolus. Eur J Drug Metab Pharmacokinet. 2013 Mar;38(1):1-4. doi: 10.1007/s13318-012-0108-7. Epub 2012 Nov 21. PMID 23179562